CLINICAL TRIAL: NCT06166485
Title: The Effect of Bath Applied in Two Different Sequences on Stress Level and Physiological Parameters in Term Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayşe Dilan Koçak, Midwife, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IstanbulUCEdu
Record Dates: First submitted 2023-10-03; First posted 2023-12-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Newborn
Keywords: baby health; stress; newborn bath; newborn

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled experimental study. Computer-assisted randomization will be used to create groups (https://www.randomizer.org/). Power analysis was performed using the G*Power (v3.1.9) program to determine the sample size. The power of the study is expressed as 1-β (β = probability of type II error) and in general, studies must have 80% power.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group babies where the head is washed first and then the whole body (Active Comparator): The effects of washing the head first and then the whole body on the physiological parameters (oxygen level, pulse, body temperature, calming time, stress level) of the first group babies will be examined.
  Interventions: Other: take a bath
- 2nd group babies, where the whole body is washed first and the head is washed last. (Active Comparator): The effects on the physiological parameters (oxygen level, pulse, body temperature, calming time, stress level) of the second group of babies, where the whole body is washed first and the head last, will be examined.
  Interventions: Other: take a bath

INTERVENTIONS:
Other: take a bath — The effects of two different bathtub bath methods on physiological parameters will be compared in babies divided into 2 different groups.

SUMMARY:
In this study, the bath applied to term babies in two different orders (first washing the body and lastly the head, and the classical method in which the whole body is washed starting from the head first), the babies' stress level, physiological parameters (body temperature, pulse, respiration, O2 saturation), procedure time (time of bathing). ) was planned to determine its effect on the calming time of babies.

The effects of two different bathing methods given to healthy and term babies on the babies' stress level, physiological parameters (body temperature, pulse, respiration, O2 saturation), procedure time (bathing time), and calming time of the babies will be compared.

DETAILED DESCRIPTION:
The researcher will briefly talk about the scope and content of the research by meeting with the parents of babies who meet the selection criteria to apply the first bath of term and healthy babies before discharge, at the earliest 6 hours after birth.

Healthy, term newborns will be divided into two groups, one group will be washed from body to head, and the other group will be washed from head to body, which is the traditional method. In the study, the stress levels of babies will be obtained by observing the newborns independently by two different observer nurses before, after and after the procedure, using the "Newborn Stress Scale", at the 5th, 15th and 30th minutes. Physiological parameters of the babies will be evaluated before the procedure, during the procedure, and at the 1st, 5th and 15th minutes after the procedure. Bathing will be done by the same person (researcher) for all babies in both the experimental and control groups.

Pulse oximeter and stopwatch will be used to measure physiological parameters (heart rate, oxygen saturation, calming time).

ELIGIBILITY:
Inclusion Criteria:

* The baby's body weight is between 2.5 - 4 kg
* The baby's Apgar score is >7
* The baby does not have any health problems
* Their parents agree to participate in the study
* Having a healthy term baby.

Exclusion Criteria:

* Meconium aspiration etc. washed immediately after birth for various reasons,
* Having various health problems,
* Their parents did not agree to participate in the study,
* Low birth weight and premature babies

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Newborn stress scale | This scale evaluation will be applied to healthy, term babies who are hospitalized in the neonatal clinic within a 3-month period and the study will be conducted.
  This scale can evaluate the stress level in newborns.Scale items are grouped into 8 subgroups.These subgroups consist of a total of 24 items in a 3-point Likert type, including facial expression, body color, respiration, activity level, consolability, muscle tone, extremities, and posture.In scoring, each subgroup is evaluated between 0-2 points. A minimum of 0 points and a maximum of 16 points are taken from the scale. As the score increases, the baby's stress level increases.
Data collection form | The 36-question data collection form will be applied to the mother of the baby on whom the study will be conducted and to the observers making the evaluation within 3 months of data collection.
  The form consists of 4 sections and 36 questions in total. The first part of the form is a 7-question form to collect demographic and obstetric information of mothers who agreed to participate in the study. The second part is a 9-question form in which information about the baby to be included in the study is collected. In the third section, it is a form with 15 questions in which information about the application is collected. In the fourth section, it is a form with 5 questions in which information regarding the evaluation of the baby with the stress scale is collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y, Zhou L, Abdillah H, Hu B, Jiang Y. Effects of swaddled and traditional tub bathing on stress and physiological parameters of preterm infants: A randomized clinical trial in China. J Pediatr Nurs. 2022 May-Jun;64:e154-e158. doi: 10.1016/j.pedn.2021.11.028. Epub 2021 Dec 23. PMID 34953663
- [Background] Kusari A, Han AM, Virgen CA, Matiz C, Rasmussen M, Friedlander SF, Eichenfield DZ. Evidence-based skin care in preterm infants. Pediatr Dermatol. 2019 Jan;36(1):16-23. doi: 10.1111/pde.13725. Epub 2018 Dec 12. PMID 30548578
- [Background] Fernandez D, Antolin-Rodriguez R. Bathing a Premature Infant in the Intensive Care Unit: A Systematic Review. J Pediatr Nurs. 2018 Sep-Oct;42:e52-e57. doi: 10.1016/j.pedn.2018.05.002. Epub 2018 May 18. PMID 29779763
- [Background] Moser WJ, Bilka KR, Vrouwe SQ, Glick JC, Ramaiah V. Running water while bathing is a risk factor for pediatric scald burns. Burns. 2023 Nov;49(7):1714-1718. doi: 10.1016/j.burns.2023.03.014. Epub 2023 Mar 23. PMID 37193613
- [Background] Ar I, Gozen D. Effects of Underrunning Water Bathing and Immersion Tub Bathing on Vital Signs of Newborn Infants: A Comparative Analysis. Adv Neonatal Care. 2018 Dec;18(6):E3-E12. doi: 10.1097/ANC.0000000000000484. PMID 30507829
- [Background] Tasdemir HI, Efe E. The effect of tub bathing and sponge bathing on neonatal comfort and physiological parameters in late preterm infants: A randomized controlled trial. Int J Nurs Stud. 2019 Nov;99:103377. doi: 10.1016/j.ijnurstu.2019.06.008. Epub 2019 Jun 21. PMID 31442786
- [Derived] Kocak AD, Inal S. The effect of bath applied in two different sequences on stress level and physiological parameters in term babies. J Pediatr Nurs. 2026 Jan 7;87:50-57. doi: 10.1016/j.pedn.2025.12.025. Online ahead of print. PMID 41505829

DOCUMENTS (3):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06166485/Prot_003.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06166485/SAP_004.pdf
  • Informed Consent Form (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06166485/ICF_005.pdf